CLINICAL TRIAL: NCT00037024
Title: Project LEAD: Promoting Health Among Populations With Early Stage Cancers
Brief Title: Study of Health Promotion in Patients With Early-Stage Breast or Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Other
Other Study IDs: Pro00009493; DUMC-1547-02-8R4ER; DUMC-1547-00-8R2ER; NCI-H02-0088; CDR0000069355
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2012-11

CONDITIONS: Breast Cancer; Depression; Fatigue; Malnutrition; Prostate Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: stage I breast cancer; stage II breast cancer; stage I prostate cancer; stage II B prostate cancer; stage II A prostate cancer; male breast cancer; fatigue; malnutrition; psychosocial effects of cancer and its treatment; depression
MeSH Terms: conditions — Breast Neoplasms; Depression; Fatigue; Malnutrition; Prostatic Neoplasms; Breast Neoplasms, Male | interventions — Therapeutics; Nutritional Support; Physical Therapy Modalities; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: fatigue assessment and management
Procedure: nutritional support
Procedure: physical therapy
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Telephone counseling by a nutritionist and a personal trainer may improve physical function and quality of life in patients who have early-stage breast cancer or prostate cancer.

PURPOSE: Randomized clinical trial to compare the effectiveness of a home-based, diet and exercise-based counseling program with that of a standard home-based counseling program in promoting health in patients who have early-stage breast cancer or prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of a diet and exercise-based home-based counseling program versus a standard home-based counseling program for improving physical function at 6 and 12 months for patients with early-stage breast or prostate cancer.
* Compare the effects of these home-based programs on diet quality, physical activity, weight status, depression, and quality of life of these patients.
* Compare the factors, such as gender, race, and social support, that interact with these home-based programs to predict program efficacy in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 arms.

* Arm I: Patients receive home-based telephone counseling by a personal nutritionist and a personal trainer.
* Arm II: Patients receive home-based standard health telephone counseling in unrelated areas of cancer care (e.g., sun exposure, screening, and falls prevention).

In both arms, counseling continues every 2 weeks for 6 months.

Patients are followed at 6 months.

PROJECTED ACCRUAL: A total of 420 patients (210 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of early-stage breast or prostate cancer within the past 18 months
* Dietary and physical activity habits and baseline functional status that places patient at risk
* Potentially able to increase physical activity and to follow a low-fat, plant-based diet
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 65 and over

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Able to speak and write English
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No other illness or condition that would preclude adherence to a plant-based diet or exercise

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 2002-04; Primary Completion 2004-02 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Demark-Wahnefried, PhD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Demark-Wahnefried W, Morey MC, Clipp EC, Pieper CF, Snyder DC, Sloane R, Cohen HJ. Leading the Way in Exercise and Diet (Project LEAD): intervening to improve function among older breast and prostate cancer survivors. Control Clin Trials. 2003 Apr;24(2):206-23. doi: 10.1016/s0197-2456(02)00266-0. PMID 12689742
- [Result] Demark-Wahnefried W, Clipp EC, Morey MC, Pieper CF, Sloane R, Snyder DC, Cohen HJ. Physical function and associations with diet and exercise: Results of a cross-sectional survey among elders with breast or prostate cancer. Int J Behav Nutr Phys Act. 2004 Oct 29;1(1):16. doi: 10.1186/1479-5868-1-16. PMID 15516261
- [Result] Demark-Wahnefried W, Clipp EC, Morey MC, Pieper CF, Sloane R, Snyder DC, Cohen HJ. Lifestyle intervention development study to improve physical function in older adults with cancer: outcomes from Project LEAD. J Clin Oncol. 2006 Jul 20;24(21):3465-73. doi: 10.1200/JCO.2006.05.7224. PMID 16849763
- [Result] Stull VB, Snyder DC, Demark-Wahnefried W. Lifestyle interventions in cancer survivors: designing programs that meet the needs of this vulnerable and growing population. J Nutr. 2007 Jan;137(1 Suppl):243S-248S. doi: 10.1093/jn/137.1.243S. PMID 17182834
- [Result] Clutter Snyder D, Sloane R, Haines PS, Miller P, Clipp EC, Morey MC, Pieper C, Cohen H, Demark-Wahnefried W. The Diet Quality Index-Revised: a tool to promote and evaluate dietary change among older cancer survivors enrolled in a home-based intervention trial. J Am Diet Assoc. 2007 Sep;107(9):1519-29. doi: 10.1016/j.jada.2007.06.014. PMID 17761229
- [Result] Morey MC, Sloane R, Pieper CF, Peterson MJ, Pearson MP, Ekelund CC, Crowley GM, Demark-Wahnefried W, Snyder DC, Clipp EC, Cohen HJ. Effect of physical activity guidelines on physical function in older adults. J Am Geriatr Soc. 2008 Oct;56(10):1873-8. doi: 10.1111/j.1532-5415.2008.01937.x. Epub 2008 Sep 17. PMID 18800990
- [Result] Demark-Wahnefried W, Morey MC, Sloane R, Snyder DC, Cohen HJ. Promoting healthy lifestyles in older cancer survivors to improve health and preserve function. J Am Geriatr Soc. 2009 Nov;57 Suppl 2(Suppl 2):S262-4. doi: 10.1111/j.1532-5415.2009.02507.x. PMID 20122025
- [Result] Morey MC, Blair CK, Sloane R, Cohen HJ, Snyder DC, Demark-Wahnefried W. Group trajectory analysis helps to identify older cancer survivors who benefit from distance-based lifestyle interventions. Cancer. 2015 Dec 15;121(24):4433-40. doi: 10.1002/cncr.29684. Epub 2015 Oct 29. PMID 26512712